CLINICAL TRIAL: NCT01382537
Title: Evaluation of the Efficacy of the InterX 5000 in the Treatment of Chronic Neck and Shoulder Pain
Brief Title: Efficacy of the InterX 5000 in the Treatment of Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Memorial Chiropractic College (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, John J Triano, Dr. John J. Triano, Canadian Memorial Chiropractic College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 072131
Record Dates: First submitted 2009-09-21; First posted 2011-06-27 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Neck Pain; Shoulder Pain
Keywords: Neck; Chronic; Musculoskeletal; Shoulder
MeSH Terms: conditions — Neck Pain; Shoulder Pain; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Device: InterX 5000
- B (Placebo Comparator)
  Interventions: Device: InterX 5000

INTERVENTIONS:
Device: InterX 5000 — A computer driven electrical stimulation unit that contains a cutaneous impedance sensor.
  Arms: A
Device: InterX 5000 — Placebo treatment
  Arms: B

SUMMARY:
This study will focus on the efficacy of treating 80 patients who have functional limitations in activity because of chronic/recurrent neck or shoulder pain.

Hypothesis 1: InterX therapy alone will have a moderate effect to reduce pain during weeks 1-2.

Hypothesis 2: Functional gains will be greater in patients receiving InterX therapy compared to those who received placebo treatment.

Hypothesis 3: Chronic neck and shoulder pain is more prevalent in patients who exhibit radiographic evidence of degenerative spondylosis/arthrosis of the cervical spine.

DETAILED DESCRIPTION:
Evaluation of subjects will be conducted at baseline (interval 0) and at 2, 4, 6 and 12 week time periods. At 26 weeks, the patient will be contacted to obtain follow-up questionnaires on pain and function. After informed consent, participants will be randomly assigned to a treatment group and a sham group using the InterX5002, hand held electrical stimulation unit. Treatment will be administered three times per week for six weeks.

During the interval of weeks 1-2 patients will have either the InterX treatment/sham alone. Weeks 3-4 will advance the patient adding a standardized rehabilitation exercise program typical for chronic neck patients. During weeks 5-6, the patient will be scheduled for treatment and will use a self-administered InterX treatment ("home" Flex) unit mimicking home care but accounting for compliance issues through attendance being monitored.

Baseline and follow-up assessments will consist of pain scores, NDI, neck fatigue testing, shoulder and arm reach tasks and walking on a treadmill at 2 MPH for 5 minutes (Neck-walk Index, NWI). Neck fatigue testing will consist of prone positioning and extensor muscle exertion against resistance to tolerance at 60% MVC. Myoelectric sensors will be taped to the skin to record muscle activity during fatigue and reach task testing. Electromagnetic sensors will be taped to a swimmers cap worn by the patient and on the skin at T1 over the spine at the shoulder level and S1 at the pelvis during the walk on the treadmill and on the shoulder and arm during reach testing.

Venipuncture will be performed at the evaluation intervals to collect blood samples for quantifying circulating inflammatory cytokines.

Analysis will focus on change in pain scores and inflammatory cytokines over the first two weeks for Hypothesis H1. Primary functional outcomes including neck fatigue and progression through neck rehabilitation exercise will be tested for Hypothesis2. The third hypothesis will be tested in two ways. First, quantification of degenerative changes (e.g.disc narrowing & osteophyte formation) on x-ray (AP & Lat screening views) will be contrasted to incidence in the published literature. Second, pain levels at baseline will be stratified into quartiles and compared to quantitative tally of degenerative changes. This data will serve as a basis for determining whether future studies using degenerative change criteria are warranted. Myoelectric activity, fatigue and head-pelvic position data will be used descriptively to assess functional differences from baseline to completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* males or females
* ages 18-65
* chronic or recurrent neck or shoulder pain
* pain of at least 3 months duration
* willing to sign consent form
* able/willing to comply with treatment schedule

Exclusion Criteria:

* age over 65 years
* clinically significant herniated disc
* spinal fracture
* previous electrical stimulation treatment for this episode
* recent cervical spine or shoulder surgery
* implanted instrumentation/prostheses
* epilepsy
* pregnancy
* recent (3 months) chemotherapy/radiotherapy
* phlebitis
* cortisone use (30 days)
* hypersensitivity to tape used with EMG

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2008-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 10 minutes
  Pain scores on the Visual Analog Scale.
Neck Disability Index | 15 minutes
  Neck Disability Index pain scores.
Shoulder Pain and Disability Index | 60 minutes
  Shoulder Pain and Disability Index scores.
Medical Outcomes Study Short-Form (SF-36) | 15 minutes
  Change in Medical Outcomes Study Short-Form (SF-36) score.
Neck Walk Index | 20 minutes
  Change in Neck Walk Index score.
Upper Limb Coordination During and Overhead Reach | 20 minutes
  Change in range of motion.
Task Limitation (TL)/Upper Limb Function - FIT-HaNSA Protocol | 20 min
  Change in FIT-HaNSA score.
EMG testing | 30 minutes
  Mean frequency shifts. Change in percentage of maximum voluntary contraction.

SECONDARY OUTCOMES:
Blood and serum biomarkers | 20 minutes
  Change in cytokine counts.

CONTACTS AND LOCATIONS:
Locations (1):
- Canadian Memorial Chiropractic College, Toronto, Ontario, Canada

REFERENCES:
- [Background] Brennan PC, Triano JJ, McGregor M, Kokjohn K, Hondras MA, Brennan DC. Enhanced neutrophil respiratory burst as a biological marker for manipulation forces: duration of the effect and association with substance P and tumor necrosis factor. J Manipulative Physiol Ther. 1992 Feb;15(2):83-9. PMID 1373431
- [Background] Godfrey CM, Morgan PP, Schatzker J. A randomized trial of manipulation for low-back pain in a medical setting. Spine (Phila Pa 1976). 1984 Apr;9(3):301-4. doi: 10.1097/00007632-198404000-00015. PMID 6233718
- [Background] Hurley DA, McDonough SM, Dempster M, Moore AP, Baxter GD. A randomized clinical trial of manipulative therapy and interferential therapy for acute low back pain. Spine (Phila Pa 1976). 2004 Oct 15;29(20):2207-16. doi: 10.1097/01.brs.0000142234.15437.da. PMID 15480130
- [Background] Pope MH, Phillips RB, Haugh LD, Hsieh CY, MacDonald L, Haldeman S. A prospective randomized three-week trial of spinal manipulation, transcutaneous muscle stimulation, massage and corset in the treatment of subacute low back pain. Spine (Phila Pa 1976). 1994 Nov 15;19(22):2571-7. doi: 10.1097/00007632-199411001-00013. PMID 7855683
- [Background] Teodorczyk-Injeyan JA, Injeyan HS, Ruegg R. Spinal manipulative therapy reduces inflammatory cytokines but not substance P production in normal subjects. J Manipulative Physiol Ther. 2006 Jan;29(1):14-21. doi: 10.1016/j.jmpt.2005.10.002. PMID 16396725
- [Derived] Teodorczyk-Injeyan JA, Triano JJ, McGregor M, Woodhouse L, Injeyan HS. Effect of Interactive Neurostimulation Therapy on Inflammatory Response in Patients With Chronic and Recurrent Mechanical Neck Pain. J Manipulative Physiol Ther. 2015 Oct;38(8):545-54. doi: 10.1016/j.jmpt.2015.08.006. Epub 2015 Oct 4. PMID 26435087